CLINICAL TRIAL: NCT05752695
Title: Risk Factors for Cruciate Ligament Injuries
Brief Title: Operation Korsband
Status: Enrolling by invitation | Type: Observational
Sponsor: Linnaeus University (Other)
Collaborators: Kalmar County Hospital (Other)
Responsible Party: Principal Investigator, Sofia Ryman Ryman Augustsson, Associate Professor, Linnaeus University
Other Study IDs: 2022-06554-01
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ACL injured athletes: Athletes with defined ACL injury.

SUMMARY:
This study aims to investigate if a detailed and comprehensive survey can identify, explain and prevent the risk factors for ACL injury.

A a new questionnaire has been developed with questions to young athletes who have suffered an anterior cruciate ligament injury. The questionnaire is more detailed and provide more information about how the anterior cruciate ligament injury occurred compared with the questionnaires currently available in the literature. This careful documentation will provide new knowledge and might be used to identify, explain and prevent risk factors that cause young athletes to suffer an anterior cruciate ligament injury.

DETAILED DESCRIPTION:
Participants will be prospectively recruited at their first physiotherapist clinical session. On this occasion, participants will be asked to fill in a questionnaire regarding injury situation, game or training, sex, age, sport affiliation, level of sport, other aspects of sport such as participation in several teams and junior versus senior games/training. In addition, questions regarding previous injury will also be documented.

ELIGIBILITY:
Inclusion Criteria:

* Athlete
* Defined ACL injury

Exclusion Criteria:

* Non athletes
* Younger than 12 years

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Athletes with ACL defined ACL injury.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Total work load | Day 1
  Total hours, per week, of practice and games.

SECONDARY OUTCOMES:
Number of teams | Day 1
  In team athletes, the number of teams in which the athlete participates.
Injury situation 1 | Day 1
  Question regarding when the injury occurred; training vs game.
Injury situation 2 | Day 1
  Question regarding at what situation the injury occurred (e.g. jump, landing, header duel, defense, attack...)
Injury situation 3 | Day 1
  Question regarding at what time, during a game, the injury occurred; approximate match minute
Physical well-being | Day 1
  Physical well-being is assessed with a likert scale ranging from 1-5 where '1' represents 'out of shape' while '5' represents that you felt 'in top shape'.
Mental wellbeing | Day 1
  Mental well-being is assessed with a likert scale ranging from 1-5 where '1' represents 'out of shape' while '5' represents that you felt 'in top shape'.
Previous injury | Day 1
  Description of previous injury prior to the ACL injury, such as other injuries to lower extremity or concussion.

CONTACTS AND LOCATIONS:
Locations (1):
- Sofia Ryman Augustsson, Kalmar, Sweden

IPD SHARING:
Plan to Share IPD: No